CLINICAL TRIAL: NCT04167046
Title: Bloc Des Muscles Erecteurs du Rachis Pour Chirurgie d'exérèse de première côte Dans le Cadre du Syndrome du défilé Cervico-thoracique: évaluation Avant-après au CHU d'Angers.
Brief Title: Erector Spinae Block in First Rib Resection: a Monocentric Before-after Study
Acronym: MERCOTE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/98
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients in this group did not receive an erector spinae block. Data are obtained retrospectively (years 2017 and 2018).
- Erector spinae block: Patients in this group receive an erector spinae block. Data will be obtained prospectively.
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: Erector spinae block — Preoperative erector spinae block.
  Groups: Erector spinae block

SUMMARY:
First rib resection surgery for thoracic outlet syndrome is associated with an intense postoperative pain. It leads to significant consumption of nonsteroidal anti-inflammatory drugs and opioids, and hospitalization for several days.

In our center, first rib resection surgery was usually performed under general anesthesia combined with diffuse local infiltration of the axillary fossa. Erector spinae block is an interfascial block where a local anesthetic is injected between the erector spinae muscle and the transverse process, in order to obtain a multimetameric analgesia. It has now shown its efficacy and its safety in thoracic and abdominal surgeries by decreasing the morphine consumption and pain scores. Since November 2018, this erector spinae block is systematically performed preoperatively for first rib resection in our center, in association with a general anesthesia. Patient satisfaction seems important but remains to be assessed objectively.

In a before-after study, our goal is to assess the impact of the use of erector spinae block on postoperative pain in the first rib resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* First rib resection for thoracic outlet syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing first rib resection for thoracic outlet syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Pain assessment at H+48 | Day 2 after surgery
  Numerical pain rating scale: 0 (no pain at all) to 10 (worst imaginable pain)

SECONDARY OUTCOMES:
Postoperative pain assessment at other times | Hour 2, Day 1, and Day 3 after surgery
  Numerical pain rating scale: 0 (no pain at all) to 10 (worst imaginable pain)
Total consumption of morphine (per and postoperative) | Hour 2, Day 1, Day 2 and Day 3 after surgery
Frequency of adverse effects related to morphine Frequency of morphine side effects | Hour 2, Day 1, Day 2 and Day 3 after surgery
Length of hospital stay | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Rineau, MD, Principal Investigator — University Hospital of Angers, France
Locations (1):
- Département d'Anesthésie-Réanimation du CHU d'Angers, Angers, France